CLINICAL TRIAL: NCT05037734
Title: A Post-Market, Multicenter, Randomized Controlled Trial of the ROSA® Partial Knee System for Unicompartmental Knee Arthroplasty
Brief Title: A Randomized Controlled Trial for Partial Knee Arthroplasty
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Relaunch at later date with updated product.
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMU2020-28CA
Record Dates: First submitted 2021-08-20; First posted 2021-09-08 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2022-05

CONDITIONS: Degenerative Joint Disease of Knee; Osteoarthritis; Traumatic Arthritis; Varus Deformity; Knee Pain Chronic
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participant will be randomized into one of the two available study arms, and will be blinded from treatment until surgery has occurred.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Robotic-Assisted UKA (Active Comparator): Randomized participant will receive UKA via the ROSA Partial Knee System.
  Interventions: Device: Persona Partial Knee System
- Traditional/Conventional UKA (Active Comparator): Randomized participant will receive the UKA via Conventional/Traditional UKA Methods.
  Interventions: Device: Persona Partial Knee System

INTERVENTIONS:
Device: Persona Partial Knee System — Unicompartmental Knee Replacement

SUMMARY:
This is a prospective, multi-center, two-arm, randomized, controlled post-market study to evaluate and compare the clinical accuracy of component placement in robotic-assisted UKA and that of traditional methods.

DETAILED DESCRIPTION:
Sites will enroll participants into two separate arms for this study (rUKA and Conventional Instrumentation), following the assigned randomization. Consecutive patients who meet all of the inclusion criteria and none of the exclusion criteria will be eligible for participation in the study and will be pre-screened for participation in the informed consent process.

The primary objective of this study is to evaluate and compare the accuracy of the ROSA® Partial Knee System in regards to implant placement with that of traditional instrumentation. This will include the assessment of the planned vs. actual component positioning.

Secondary Objectives include the evaluation of safety and efficacy of this system and will include the assessment of common adverse events, physical exam findings, radiologic results and patient reported outcome measures.

Data collection will occur at the following intervals: Pre-operative, Operative, 6-weeks, 3-months, 1-year, and 2-years. Enrollment for the study is anticipated to last approximately 12-18 months. Allowing for 24 months of follow-up, the total estimated study time to final-patient final-visit will be approximately 42 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patient meets the approved indications for use in accordance with product labeling for both the Persona Partial Knee System and the ROSA® Partial Knee System.
2. Body mass index ≤40 kg/m2
3. Patient is of legal age and skeletally mature
4. Patient is willing and able to provide informed consent.
5. Patient is willing to be randomized into one of two study groups of UKA performed using ROSA® and UKA using Conventional Instrumentation
6. Patient is willing and able to complete scheduled follow-up evaluations as defined in the study protocol.
7. Patient qualifies for primary UKA based on investigator's clinical judgement and has an intact anterior cruciate ligament.
8. Independent of study participation, patient is a candidate for the commercially available Persona Partial Knee System.

Exclusion Criteria:

1. Independent of study participation, patient meets any of the contraindications for use in accordance with product labeling of the Persona Partial Knee System and/or the ROSA® Partial Knee System.
2. Orthopaedic procedure or pain management study of any joint within the last or next 6 months; furthermore, bilateral enrollment is excluded in this study.
3. Prior ACL Repair
4. Moderate to severe patello-femoral arthritis, that in the opinion of the investigator, would require patella-femoral arthroplasty.
5. Patient is unwilling to sign the Informed Consent.
6. Would, in the investigator's opinion, be unwilling or unable to comply with the postoperative care instructions or study follow-up schedule.
7. Patient is considered a member of a protected/vulnerable population (Pregnant, prisoner, mentally incompetent, etc.).
8. Patient is institutionalized or is a known drug abuser, a known alcoholic or cannot understand the requirements of study participation.
9. Patient has a condition which would, in the judgement of the investigator, place the patient at undue risk or interfere with the conduct of the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06 (Estimated); Primary Completion 2030-06 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy of implant position | 6 Weeks
  To compare and evaluate the accuracy of implant position of robotic-arm surgical assistant (ROSA® Partial Knee System) with that of conventional instrumentation (Traditional UKA). Accuracy of the Implemented Plan will be evaluated by assessing Implant alignment post-operatively for participants enrolled for both Conventional Instrumentation and the ROSA® Partial Knee System.

SECONDARY OUTCOMES:
Evaluation of Patient safety | 24 months
  Frequency and incidence of adverse events, serious adverse events, adverse device effects, serious adverse device effects, and unanticipated serious adverse device effects as well as device deficiencies.
Evaluation of range of motion | 24 months
  Evaluation of knee flexion/extension pre-operatively and post-operatively
Evaluation of Instability | 24 months
  Medial/Lateral and Anterior/Posterior instability measured from none to severe(>5mm).
Patient Reported Outcome Measure (Oxford Knee Score) | 24 months
  A questionnaire completed by the patient consisting of twelve questions that utilize a 5-point Likert scoring system (0 - 4) resulting in a score ranging from 0 (worst) to 48 (best).
Patient Reported Outcome Measure (KOOS-12) | 24 months
  A questionnaire completed by the patient consisting of a 12-item short form of the original 42-item Knee Injury Osteoarthritis Outcome Score (KOOS), and will be used to measure the patients' perception of pain, function, and knee-related quality of life
Numeric Pain Rating Scale (NPRS) | 24 Months
  An 11-point NPRS is a patient self-completed reported outcome and will be used to assess the current level of pain for the affected hip. On this scale, 0 will indicate no pain and 10 will indicate the worst pain imaginable
Subject Satisfaction | 24 Months
  A questionnaire consisting of a single satisfaction question in regard to the subjects knee replacement. Answers will include the following: Very Dissatisfied, Dissatisfied, Neutral, Satisfied, Very Satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Hillary Overholser, Study Director — Zimmer Biomet
Locations (1):
- Mississippi Sports Medicine and Orthopaedic Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No